CLINICAL TRIAL: NCT02571686
Title: Accuracy of Pulse Oximeters With Profound Hypoxia
Status: Completed | Type: Observational
Sponsor: Mortara Instrument (Industry)
Responsible Party: Sponsor
Other Study IDs: 139253
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Oximetry, Pulse

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Surveyor S4

SUMMARY:
The aim of this project is to test the accuracy of pulse oximeters during mild, moderate and severe hypoxia. This is done by comparing the reading of the pulse oximeter during brief, steady state hypoxia with a gold-standard measurement of blood oxyhemoglobin saturation (arterial blood sample processed in a laboratory hemoximeter). The data obtained is submitted by pulse oximeter manufacturers to the FDA for device approval.

DETAILED DESCRIPTION:
Overall design:

Studies normally involve 6-12 normal adult volunteer paid subjects, with 20-25 1-2 ml arterial blood samples from each subject obtained at different steady-state levels of hypoxia from 70-100%. Blood samples obtained from an arterial line are measured in a hemoximeter to determine true saturation value. Some sponsors may not require any blood sampling. Some sponsors may require additional blood samples, up to 35 samples may be drawn.

Readings from the test pulse oximeters are recorded and compared to these "gold-standard" blood values. The pulse oximeter probes may be located at a variety of sites on the subjects, including fingers, toes, ears, forehead, scalp and bridge of the nose. These detector-probes are all non-invasive. The level of hypoxia is measured and controlled by the investigator. A computer program that displays a prediction, breath by breath, the arterial oxygen saturation, (SaO2) of the study subject. SaO2 is computed from end-expired Po2 and Pco2 as determined by mass spectrometer gas analysis. This information permits the inspired gas mixture of air, plus CO2 and nitrogen, to be adjusted by an operator watching the value computed after each expiration on an analog meter. This computer-estimated saturation is adjusted by the operator to one of 6 levels of predicted saturation, and is held stable for about 30 seconds at each level. Two or three "runs" are conducted per subject. Each "run" lasts 8-12 min and 4 to 5 plateaus are tested per run. The manufacturer may choose the target values. Plateaus are typically sought at 92%, 86%, 80%, 74%, 68% and 62%. Other manufacturers have asked for an equal number of data points but with all points between 70% and 100%. Some sponsors may also request additional variables to be measured during testing including high or low Carbon Dioxide (CO2), where subjects will be asked to hyperventilate; low perfusion, where subjects will be asked to lay flat, or with their head up or down; testing pulse oximeters during motion, with the subject's hand fixed to a motion machine; or measure eye-tracking during hypoxia. The subject's will be informed by the study staff and in the consent form if any of these additional procedures apply.

.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female, aged ≥18 and <50.
2. The subject is in good general health with no evidence of any medical problems.
3. The subject is fluent in both written and spoken English.
4. The subject has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

1. The subject is obese (BMI>30).
2. The subject has a known history of heart disease, lung disease, kidney or liver disease.
3. Diagnosis of asthma, sleep apnea, or use of CPAP(Continuous positive airway pressure).
4. Subject has diabetes.
5. Subject has a clotting disorder.
6. The subject a hemoglobinopathy or history of anemia, per subject report or the first blood sample, that in the opinion of the investigator, would make them unsuitable for study participation.
7. The subject has any other serious systemic illness.
8. The subject is a current smoker.
9. Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators' would interfere with the sensors working correctly.
10. The subject has a history of fainting or vasovagal response.
11. The subject has a history of sensitivity to local anesthesia.
12. The subject has a diagnosis of Raynaud's disease.
13. The subject has unacceptable collateral circulation based on exam by the investigator (Allen's test).
14. The subject is pregnant, lactating or trying to get pregnant.
15. The subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures.
16. The subject has any other condition, which in the opinion of the investigators' would make them unsuitable for the study -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 10-12 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Accuracy of Pulse Oximeter | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia Clinical Studies Facility, room A-65 Parnassus Campus., San Francisco, California, United States